CLINICAL TRIAL: NCT03795038
Title: Comparison of the Plasma Lipoprotein Apheresis Systems DIAMED and MONET vs. the Whole Blood Apheresis System DALI: Cross-over Study in Patients With Cardiovascular Disease and Severe Dyslipidemia
Brief Title: Comparison of the Plasma Lipoprotein Apheresis Systems DIAMED and MONET vs. the Whole Blood Apheresis System DALI
Acronym: DIAMOND-2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TA-DMD-01-D
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Hypercholesterolemia, Familial; Dyslipidemias; Cardiovascular Diseases
Keywords: Lipoprotein apheresis
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Dyslipidemias; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, open, interventional, cross-over with randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipoprotein Apheresis MONET and DALI (Other): Patients routinely treated with MONET:
  * The first subgroup will be treated first with the MONET adsorber system for three consecutive treatments followed by a treatment for three consecutive treatments with the DALI adsorber System.
  * The second subgroup will be treated first with the DALI adsorber system for three consecutive treatments followed by a treatment for three consecutive treatments with the MONET adsorber system
  Interventions: Device: Lipoprotein Apheresis MONET and DALI
- Lipoprotein Apheresis DIAMED and DALI (Other): Patients routinely treated with DIAMED:
  * The first subgroup will be treated first with the DIAMED adsorber system for three consecutive treatments followed by a treatment for three consecutive treatments with the DALI adsorber system.
  * The second subgroup will be treated first with the DALI adsorber system for three consecutive treatments followed by a treatment for three consecutive treatments with the DIAMED adsorber System.
  Interventions: Device: Lipoprotein Apheresis DIAMED and DALI

INTERVENTIONS:
Device: Lipoprotein Apheresis MONET and DALI — Three apheresis treatments assigned to one type of apheresis system of MONETand DALI
  Arms: Lipoprotein Apheresis MONET and DALI
Device: Lipoprotein Apheresis DIAMED and DALI — Three apheresis treatments assigned to one type of apheresis system of DIAMOND and DALI
  Arms: Lipoprotein Apheresis DIAMED and DALI

SUMMARY:
The clinical Investigation will be performed to compare the safety and effectiveness of the CE certified and established lipoprotein apheresis systems MONET vs. DALI and DIAMED vs. DALI for optimizing the individual therapy of patients with severe dyslipidemia using established and novel efficacy parameters.

DETAILED DESCRIPTION:
Comparison of the safety and effectiveness of the CE certified and established lipoprotein apheresis systems MONET vs. DALI and DIAMED vs. DALI for optimizing the individual therapy of patients with severe dyslipidemia using established and novel efficacy parameters.

The primary objective is to compare the whole blood lipoprotein apheresis system DALI with the plasma lipoprotein apheresis systems MONET and DIAMED with regard to their efficacies in removing total cholesterol, low density lipoprotein cholesterol (LDL-C), triglycerides and lipoprotein (a) (Lp(a)).

The secondary objective is to compare the whole blood lipoprotein apheresis system DALI with the plasma lipoprotein apheresis system MONET and DIAMED with regard to their efficacies in removing other novel efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by study patient and investigator/authorised physician
* Minimum age of 18 years
* Ability to understand the nature and requirements of the study

Study-specific inclusion criteria:

* Patients with indication for lipoprotein apheresis confirmed by a local apheresis expert commission according to the German guidelines [1] and with routine lipoprotein apheresis treatments for at least 3 months. Patients with weekly treatments have not missed more than 3 treatment sessions within the 3 months prior inclusion to the study. Patients with biweekly treatment sessions have not missed more than 1 treatment session within the 3 months prior inclusion to the study
* Patients with regular weekly or biweekly lipoprotein apheresis treatments with either MONET or DIAMED lipoprotein apheresis systems for at least 4 weeks (weekly treatments) or 8 weeks (biweekly treatments) with the same system
* With adequate venous access
* With systolic blood pressure > 100 mmHg
* With stable hematocrit >35 %
* With stable anticoagulation

Exclusion Criteria:

* Any condition which could interfere with the patient's ability to comply with the study
* Pregnancy or lactation period (pregnancy test will be conducted with female patients aged 55 years)
* Participation in an interventional clinical study during the preceding 30 days or in the same study

Study-specific exclusion criteria:

* Occurrence or clinical relevant deterioration of acute myocardial infarction, unstable angina pectoris, severe hemo-dynamic relevant arrhythmia within 3 months prior inclusion to the study
* Bypass surgery, vascular diseases, active infection (this means chronic infectious diseases (e.g. chronic hepatitis) and acute infections with a core body temperature ≥ 38.0 °C) or unstable circulation (see exclusion criteria no. 7) within the last 3 months
* Uncontrolled high or low blood pressure defined as systolic blood pressure >180 mmHg/<100 mmHg and/or diastolic blood pressure >115 mmHg (after three times measuring)
* Changes in lipid lowering medication within the last 2 weeks
* Intake of Angiotensin Converting Enzyme (ACE) inhibitor medication within a time interval of five times the terminal half-life of the ACE inhibitor before study start and during the study
* History of allergic reactions to anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Removal rate of total cholesterol | every week for 6 weeks or biweekly for 12 weeks
  Removal rate of total cholesterol as primary endpoint in blood samples to evaluate the clinical performance of the apheresis systems
Removal rate of low density lipoprotein cholesterol (LDL-C) | every week for 6 weeks or biweekly for 12 weeks
  Removal rate of low density lipoprotein cholesterol (LDL-C) as primary endpoint in blood samples to evaluate the clinical performance of the apheresis systems
Removal rate of triglycerides | every week for 6 weeks or biweekly for 12 weeks
  Removal rate of triglycerides as primary endpoint in blood samples to evaluate the clinical performance of the apheresis systems
Removal rate of lipoprotein (a) (Lp(a)). | every week for 6 weeks or biweekly for 12 weeks
  Removal rate of lipoprotein (a) (Lp(a)) as primary endpoint in blood samples to evaluate the clinical performance of the apheresis systems

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Prophet, Dr. med., Principal Investigator — Nephrocare Rostock GmbH
Locations (2):
- Germany (2):
  - Nephrocare Rostock GmbH, Rostock, Mecklenburg-Vorpommern
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony